CLINICAL TRIAL: NCT03564587
Title: Improving Health-Promoting Behaviors in Adolescent Cancer Survivors Using AWAKE: A Feasibility Trial
Acronym: CHOA AWAKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Karen Effinger, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099050
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Health Behavior
Keywords: Cancer Survivors; Adolescent; Achieving Wellness After Kancer in Early Life; AWAKE; Health-Promoting Behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWAKE (Experimental): The AWAKE intervention is an 8 week program including a mobile app and phone-based coaching, focused on improving hope in order to increase quality of life and health-promoting behaviors in young adult cancer survivors.
  Interventions: Behavioral: AWAKE
- No treatment (No Intervention): Control participants will receive the surveys to complete only; however, they may opt to receive the intervention after the 4-month assessment.

INTERVENTIONS:
Behavioral: AWAKE — Behavioral intervention called Achieving Wellness After Kancer in Early Life (AWAKE) is focused on increasing hope in order to improve quality of life and health-promoting behaviors in survivors of young adult cancer. The AWAKE mobile app contains eight modules for participants to complete over 8 weeks with the ability to review prior modules. Participants receive a prompt on their mobile device weekly to complete each module and/or they will receive a text reminder. The app includes health education messaging, weekly homework assignments, the ability to track progress towards goals with self-monitoring and graphical depictions of progress, videos of inspirational materials, and a portal for interacting with their coach.
  Arms: AWAKE

SUMMARY:
A behavioral intervention called Achieving Wellness After Kancer in Early Life (AWAKE) focused on increasing hope in order to improve quality of life and health-promoting behaviors in survivors of young adult cancer. The goals of this project are to adapt the AWAKE platform into an intervention acceptable for use in adolescent cancer survivors and their guardians in order to improve survivors' hope, quality of life, and health-promoting behaviors, and to generate the preliminary data needed for a randomized control trial to test the efficacy of the AWAKE platform in this population.

DETAILED DESCRIPTION:
A behavioral intervention called Achieving Wellness After Kancer in Early Life (AWAKE) focused on increasing hope in order to improve quality of life and health-promoting behaviors in survivors of young adult cancer. Adaptation of this intervention to incorporate messaging for adolescents and their guardians has the potential to have a long-term impact on adolescent cancer survivors. The goals of this project are to adapt the AWAKE platform into an intervention acceptable for use in adolescent cancer survivors and their guardians in order to improve survivors' hope, quality of life, and health-promoting behaviors, and to generate the preliminary data needed for a randomized control trial to test the efficacy of the AWAKE platform in this population.

ELIGIBILITY:
Inclusion Criteria:

Adolescent survivors:

* Early survivor: 3 months to 2 years after therapy completion
* Long-term survivor: ≥2 years after therapy completion
* 13-17 years of age
* Access to tablet or smartphone and internet

One designated guardian per survivor

Exclusion Criteria:

* Cognitive delay that would preclude participation
* Participant or designated guardian unable to read English
* Active disease relapse

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in the he Children's Hope Scale score | Baseline, 2 and 4 months follow up visits
  A 6-item self-report questionnaire assessing children's dispositional hope. Two components, agency (ability to initiate and sustain action towards goals) and pathways (capacity to find a means to carry out goals), are assessed by the measure. Responses are on a 6-point Likert-scale ranging from 1=none of the time to 6=all of the time with higher scores representing increased dispositional hope.

SECONDARY OUTCOMES:
Change in the Pediatric Quality of Life Inventory (PedsQL), 4.0 scale score | Baseline, 2 and 4 months follow up visits
  The PedsQL 4.0 scale has 23-items that are grouped into four domains: 1)Physical Functioning (eight items), 2) Emotional Functioning (five items), 3) Social Functioning (five items) and 4) School Functioning (five items). 5-point response scale is utilized across child self-report and parent proxy-report (0 never a problem; 1 almost never a problem; 2 sometimes a problem; 3 often a problem; 4 almost always a problem). Subjects are requested to rate how much problems they experienced during the past month. All items are reverse-scored and linearly transformed to a 0 100 scale (0 100, 1 75, 2 50, 3 25, 4 0), so that higher scores indicate better Health-related quality of life (HRQoL).
Change in number of servings of fruits and vegetables | Baseline, 2 and 4 months follow up visits
  Change in number of servings of fruits and vegetables will be assessed using 9 dietary habits questions from Risk Behavior Surveillance System (YRBSS) survey
Change in number of physical activity hours per day | Baseline, 2 and 4 months follow up visits
  Change in number of physical activity hours per day will be assessed using 5 physical activity questions from Risk Behavior Surveillance System (YRBSS) survey
Change in number of screen time hours per day | Baseline, 2 and 4 months follow up visits
  Change in number of screen time hours per day will be will be assessed using a question from Risk Behavior Surveillance System (YRBSS) survey
Change in PROMIS score | Baseline, 2 and 4 months follow up visits
  The PROMIS Peer Relationships, Anxiety, and Depression scales have self-report and parent-proxy versions. Each scale is scored from 0-100 with higher scores indicating better peer relationships, worse anxiety and worse depression. Questions: 8 peer relationships, 8 anxiety, 8 depression
Usability of AWAKE | 2 month assessment
  Responses to four usability questions will be based on a 5-point Likert scale (1=very useless/ineffective; 5=very useful/effective) with higher ratings indicating more favorable attitudes.
Satisfaction with AWAKE | 2 month assessment
  Responses to 16 satisfaction questions will be based on a 5-point Likert scale (1=very useless/ineffective; 5=very useful/effective) with higher ratings indicating more favorable attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Effinger, MD, MS, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States